CLINICAL TRIAL: NCT03833557
Title: Success Rate of Three Capping Materials Used in Pulpotomy of Primary Molars: A Randomized Clinical Trial
Brief Title: Success Rate of Three Capping Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Youssef Abd Al Gawad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 181053
Record Dates: First submitted 2019-01-30; First posted 2019-02-07 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Caries
Keywords: Formocresol; MTA; Nanohydroxyapatite; Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nanohydroxyapatite Pulpotomy (Active Comparator): Biphasic calcium phosphate. Straumann BoneCeramic Regenerative Pulpotomy of 24 mandibular second primary molars using Nanohydroxyapatite
  In Group 1: 24 mandibular second primary molars Caries removal and deroofing of pulp chamber Following the manufacturer's instructions, Nanohydroxyapatite was mixed with distilled water to homogeneous consistency then introduced into the pulp chamber and condensed properly against the pulp orifices.
  All Molars were finally restored with stainless steel crowns cemented with GI cement . An immediate postoperative radiograph using periapical film size two was taken.
  Clinical and radiographic evaluation: All treated patients were followed up at one, three , six & 12 months after the pulpotomy
  Interventions: Procedure: Nanohydroxyapatite Pulpotomy
- MTA Pulpotomy (Active Comparator): Angelus Grey MTA , Regenerative Pulpotomy Pulpotomy of 24 mandibular second primary molars using MTA Caries removal and deroofing of pulp chamber The MTA powder was mixed with sterile water in a 3:1 powder/water ratio according to the manufacturer's instructions to obtain a thick creamy paste, then placed on the floor of the pulp chamber using a messing gun and compacted against the pulp orifices with a condenser over a moist cotton pellet.
  All Molars were finally restored with stainless steel crowns cemented with GI cement . An immediate postoperative radiograph using periapical film size two was taken.
  Clinical and radiographic evaluation at one, three ,six & 12 months after pulpotomy.
  Interventions: Procedure: MTA pulpotomy
- Formocresl Pulpotomy (Active Comparator): Buckley' s Formocresol , Fixation pulpotomy Pulpotomy of 24 mandibular second primary molars using Formocresol Caries removal and deroofing of pulp chamber
  A cotton pellet with formocresol was placed on the pulp stumps then removed and ZO/E dressing was condensed against the pulp stumps.
  All Molars were finally restored with stainless steel crowns cemented with GI cement . An immediate postoperative radiograph using periapical film size two was taken.
  Clinical and radiographic evaluation: All treated patients were followed up at one, three , six & 12 months after the pulpotomy for clinical and radiographic evaluation. Independently, two examiners evaluated the teeth clinically and radiographically.
  Interventions: Procedure: Formocresol Pulpotomy

INTERVENTIONS:
Procedure: Nanohydroxyapatite Pulpotomy — Biphasic calcium phosphate 500-1000 Um Straumann BoneCeramic
  Arms: Nanohydroxyapatite Pulpotomy
Procedure: MTA pulpotomy — Angleus grey MTA
  Arms: MTA Pulpotomy
Procedure: Formocresol Pulpotomy — Buckley's Fromocresol. diluted full strength foromocresol
  Arms: Formocresl Pulpotomy

SUMMARY:
A randomized clinical trial was carried out on 72 second primary molars indicated for pulpotomy divided into three equal groups (n=24) . First group received Nanohydroxyapatite as a pulpotomy agent , second group received Mineral Trioxide Aggregate ( MTA) & the third received Formocresol pulpotomy. All pulpotomized teeth were finally restored with stainless steel crowns. Subjects were monitored clinically and radiographically at one, three , six & 12 months.

DETAILED DESCRIPTION:
The study population included four to eight years old healthy and cooperative patients who presented at the Pediatric Dental Clinic, Faculty of Dentistry, Cairo University with mandibular second primary molars indicated for pulpotomy which met specific inclusion and exclusion criteria. Written consent was obtained from the parent/guardian after explaining the full details of the treatment procedure.

Procedures:

Preoperative periapical radiograph using periapical film size two Speed D Film , was taken for the molars considered for treatment. Radiographs should be of proper film density and contrast for proper radiographic diagnosis.

The pulpotomy procedure was performed by the same operator. Local anesthesia was induced and rubber dam isolation was performed, followed by caries removal and deroofing of the pulp chamber using a #330 high-speed carbide bur mounted in a water-cooled high speed turbine. The coronal pulp tissue was amputated using a sterile sharp spoon excavator. The pulp chamber was irrigated with physiologic saline. Pulp homeostasis was achieved using a sterile wet cotton pellet applied for two to three min.

In Group 1:

Following the manufacturer's instructions, Nanohydroxyapatite was mixed with distilled water to homogeneous consistency then introduced into the pulp chamber and condensed properly against the pulp orifices.

In Group 2:

The MTA powder was mixed with sterile water in a 3:1 powder/water ratio according to the manufacturer's instructions to obtain a thick creamy paste, then placed on the floor of the pulp chamber using a messing gun and compacted against the pulp orifices with a condenser over a moist cotton pellet.

Group 3:

A cotton pellet with formocresol was placed on the pulp stumps then removed and ZO/E dressing was condensed against the pulp stumps.

All Molars were finally restored with stainless steel crowns cemented with GI cement . An immediate postoperative radiograph using periapical film size two was taken.

Clinical and radiographic evaluation:

All treated patients were followed up at one, three , six & 12 months after the pulpotomy.

The pulpotomized teeth were judged as clinically successful if they met the following criteria: Absence of sensitivity, pain, tenderness to percussion, abscess, fistula or tooth mobility. Radiographic success was defined if there were normal periodontal ligament space, absence of furcation or periapical radiolucency, absence of internal or external root resorption

Statistical analysis:

Data were collected, revised for completeness and logical consistency, tabulated, and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Absence of tenderness to percussion.

  * Absence of physiologic or pathologic tooth mobility.
  * No clinical evidence of pulpal inflammation or degeneration, such as history of swelling or presence of sinus tract.
  * Restorable teeth.
  * Absence of radiographic evidence of internal or external root resorption, pulpal calcification, or osseous disease (periapical or furcation infection

Exclusion Criteria:

* • Evidence of necrosis after access cavity preparation.

  * Hemostasis could not be achieved within three min after direct contact with a wet cotton pellet, prior to material placement.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 12 Month
  abscence of all clinical signs and symptoms of failure

SECONDARY OUTCOMES:
Radiographic success rate | 12 Month
  Absence of any radiographic signs of failure

CONTACTS AND LOCATIONS:
Locations (1):
- Randa Youssef, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study design and procedures
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Abd Al Gawad RY, Hanafy RMH. Success rate of three capping materials used in pulpotomy of primary molars: A randomized clinical trial. Saudi Dent J. 2021 Nov;33(7):560-567. doi: 10.1016/j.sdentj.2020.08.007. Epub 2020 Aug 29. PMID 34803301